CLINICAL TRIAL: NCT06623461
Title: A Phase II Randomized Trial of LND101 for Fecal Microbiota Transplantation in Combination With Immune Checkpoint Blockade in Patients With Advanced Melanoma
Brief Title: LND101 for Fecal Microbiota Transplantation in Combination With Immune Checkpoint Blockade in Advanced Melanoma
Acronym: Canbiome2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Cancer Society (CCS) (Other); Weston Family Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ME17
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care ICB (Active Comparator): Assigned single agent or combination ICB treatment
  Interventions: Drug: Standard of Care Immune Checkpoint Blockade
- LND101 for FMT + Standard-of-care ICB (Experimental): Bowel preparation; LND101(single-dose); Assigned single agent or combination ICB treatment.
  Interventions: Drug: Standard of Care Immune Checkpoint Blockade; Drug: LND101

INTERVENTIONS:
Drug: Standard of Care Immune Checkpoint Blockade — Any ICB (single agent or combination) may be used that is commercially available, Health Canada-approved and publically funded for the treatment of participants with advanced, unresectable or metastatic melanoma. The treatment decision for choice of ICB regimen will be made prior to randomization and cannot be changed after enrollment
Drug: LND101 — Approximately 40 capsules (total of 80-100g of processed fecal material) taken by mouth 7 days prior to the ICG agent(s) administered following bowel preparation.
  Arms: LND101 for FMT + Standard-of-care ICB

SUMMARY:
This study is being done to answer the following question: Can the chance of melanoma growing or spreading be lowered by receiving a treatment called LND101 for Fecal Microbiota Transplant (FMT) in addition to the usual immunotherapy treatment called Immune Checkpoint Blockade (ICB)? FMT treatment changes the bacteria in your gut called the microbiome.

DETAILED DESCRIPTION:
We are doing this study because we want to find out if this approach (adding LND101 FMT to ICB) is better or worse than the usual approach (ICB only) for advanced melanoma. The usual approach is defined as care most people get for advanced melanoma.

The usual approach for patients who are not in a study is treatment with immunotherapy drugs called immune checkpoint blockade (ICB) drugs. Immunotherapy works by activating the immune system to target the cancer. This may help to slow down the growth of cancer and may cause cancer cells to die.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed histological diagnosis of cutaneous melanoma or melanoma of unknown primary.
* Participants must have stage IV or advanced unresectable disease.
* No prior ICB treatment for advanced unresectable or metastatic disease. Participants may have received adjuvant or neoadjuvant ICB if last dose was given ≥ 6 months prior to enrollment
* Prior targeted therapy with BRAF/MEK inhibition in the adjuvant or advanced / metastatic setting is permitted if at least 2 weeks have elapsed between the last dose and study enrollment. Participants must have recovered to ≤ grade 1 from all toxicity related to BRAF/MEK inhibition
* Prior radiation therapy is permitted if at least 7 days have elapsed between the last fraction and study enrollment. Participants must have recovered to ≤ grade 1 from all toxicity related to prior radiotherapy.
* Previous major surgery is permitted provided that surgery occurred ≥ 14 days prior to participant enrollment and that wound healing has occurred.
* Participants must have measurable disease as per RECIST 1.1/ iRECIST.
* Participants must be at least 18 years of age.
* Participants must have an ECOG performance status of 0, 1, or 2.
* The participant's standard-of-care ICB regimen must be selected prior to enrollment and must stay the same, regardless of arm assignment, post-enrollment
* Participants must demonstrate adequate organ function Participants must be able to ingest capsules.
* Participants must consent to provision of samples of blood and stool for correlative marker analysis.
* Participants must consent to provision of, and investigator must agree to submit, a representative archival formalin fixed paraffin block of tumour tissue for correlative analyses when tumour tissue is available.
* Participants must have access to provincially-funded standard-of-care ICB treatment.
* Participant consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each participant must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Participants must be accessible for treatment and follow-up. Investigators must assure themselves the participants randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* Protocol ICB treatment must begin within 14 calendar days after participant enrollment.
* Participants of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion Criteria:

* Participants with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Participants who have received antibiotics within 14 days of enrollment.
* Participants with systemic prednisone use > 10mg per day or equivalent dose.
* Participants with concurrent treatment with other anti-cancer therapy.
* Participants that have received live attenuated vaccination administered within 30 days prior to randomization. Note: Seasonal vaccines for influenza and COVID-19 are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and not allowed.
* For participants with history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with absolute contraindications to FMT including: a) Toxic megacolon; b) Inflammatory bowel disease; c) Severe dietary allergies
* Participants with hypersensitivity to PegLyte®
* Participants with symptomatic brain metastases unless brain lesions are shown to be stable, according to the following definitions:

  1. without evidence of progression for at least four weeks prior to randomization and have no evidence of new or enlarging brain metastases; or
  2. treated with surgery and without evidence of progression prior to randomization and have no evidence of new or enlarging brain metastases; or
  3. treated with stereotactic radiosurgery and without evidence of progression prior to randomization and have no evidence of new or enlarging brain metastases.
  4. asymptomatic or minimally symptomatic active metastases, with controlled steriod use and no imminent CNS complications.
* Participants with leptomeningeal disease.
* Participants with any uncontrolled autoimmune disease that requires active immunosuppressive agents.
* Participants who are solid organ transplantation recipients or likely to receive solid organ transplants in the future.
* Participants living with HIV.
* Participants with active infection. Participants may be eligible following recovery. Participants requiring antibiotics require 2-week washout period prior to enrollment.
* Participants that are pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 4 years

SECONDARY OUTCOMES:
Overall Survival | 4 years
Objective Response Rate | 4 years
Number and severity of adverse events assessed with CTCAE version 5.0 | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Elkrief, Study Chair — CHUM-Centre Hospitalier de ''Universite de Montreal, Montreal, QC Canada; John Lenehan, Study Chair — London Regional Cancer Program, London, ON Canada
Locations (14):
- Canada (14):
  - BCCA - Abbotsford, Abbotsford, British Columbia
  - BCCA - Surrey, Surrey, British Columbia
  - BCCA - Vancouver, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre Research Inc., London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Centre Integre de Sante et de Services Sociaux, Greenfield Park, Quebec
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec
  - Centre hospitalier regional de Trois-Rivieres, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: Yes
As per CCTG policies.
URL: https://www.ctg.queensu.ca/public/policies

REFERENCES:
- [Derived] Hadi DK, Baines KJ, Jabbarizadeh B, Miller WH, Jamal R, Ernst S, Logan D, Belanger K, Esfahani K, Elkrief A, Parvathy SN, Silverman MS, Routy B, Maleki Vareki S, Lenehan JG. Improved survival in advanced melanoma patients treated with fecal microbiota transplantation using healthy donor stool in combination with anti-PD1: final results of the MIMic phase 1 trial. J Immunother Cancer. 2025 Aug 4;13(8):e012659. doi: 10.1136/jitc-2025-012659. PMID 40759441